CLINICAL TRIAL: NCT00225420
Title: A Phase I/II Study of Concurrent Weekly Docetaxel (Taxotere®), Androgen Ablation, and Adaptive External Beam Radiotherapy for Localized High-Risk Adenocarcinoma of the Prostate
Brief Title: Docetaxel, Androgen Ablation, and External-Beam Radiation Therapy in Patients With High-Risk Localized Prostate Cancer
Acronym: NRR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0420
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Leuprolide; luprolide acetate gel depot; Goserelin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Intervention (Other): Single Arm Intervention where after enrollment (or prior to enrollment but before starting radiotherapy) patients will initially receive leuprolide acetate (Lupron®) intramuscular (IM). Patients will begin adaptive external-beam radiation therapy 2-3 months following the initiation of hormonal therapy. Each patient receives a dose of docetaxel at 10 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight weeks.
  Interventions: Drug: docetaxel; Drug: leuprolide acetate; Radiation: radiation therapy

INTERVENTIONS:
Drug: docetaxel — Docetaxel will be administered per the designated cohort starting at 10 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  Other Names: Taxotere
Drug: leuprolide acetate — Leuprolide acetate will be administered at 22.5 mg IM and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  Other Names: Lupron; Eligard; Viadur; Zoladex
Radiation: radiation therapy — The total dose will be 7800 cGy in 200 centigray (cGy) per fraction for a total of 39 treatments.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide, may lessen the amount of androgens made by the body. Radiation therapy uses high energy x-rays to kill tumor cells. Giving docetaxel together with androgen ablation therapy and external-beam radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of docetaxel when given together with androgen ablation therapy and external-beam radiation therapy and to see how well they work in treating patients with high-risk localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of docetaxel when administered in combination with androgen ablation therapy and adaptive external-beam radiotherapy in patients with high-risk localized adenocarcinoma of the prostate.

Secondary

* Determine the 2-year biochemical progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter, open-label, dose-escalation study of docetaxel.

* Androgen ablation therapy: Patients receive leuprolide acetate or other luteinizing hormone-releasing hormone agonist beginning 2-3 months prior to the start of chemoradiotherapy and continuing for up to 2 years.
* Chemoradiotherapy: Patients receive docetaxel IV over 1 hour on day 1 and high-dose external-beam radiotherapy on days 1-5. Treatment repeats every 7 days for 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate with any of following clinical features:

   A) T3 or T4 B) T1-2 + Gleason Score 8-10 C) T1-2 + Gleason Score 7 + Prostate Specific Antigen (PSA) >10 ng/mL D) T1-2 + Any Gleason Score + PSA >20 ng/mL
2. No evidence of metastatic disease on chest x-ray, bone scan or CT scan of abdomen/pelvis.
3. Age > 18
4. The Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
5. Peripheral neuropathy: must be < grade 1
6. Hematologic parameters A) Absolute neutrophil count > 1,500/mm3 B) Hemoglobin > 8.0 g/dL C) Platelet count > 100,000/mm3.
7. Hepatic parameters / Renal function A) Total Bilirubin must be ≤ 1.2 mg/dL B) Transaminases (AST and ALT) must be < 1.5 x upper limit of normal (ULN) C) Alkaline phosphatase must be < 2.5 x ULN D) Creatinine < 1.5 x ULN ( < 2.1 mg/dL)
8. No prior pelvic or prostate radiation or chemotherapy for prostate cancer. Androgen ablation therapy with one of the luteinizing hormone-releasing hormone (LH-RH) agonists prior to enrollment is acceptable as long as protocol treatment with radiotherapy and chemotherapy is started within 3 months of the initiation of androgen ablation.
9. Patient must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

1. Documented metastases on staging studies
2. Life expectancy <10 years secondary to co-morbid illness
3. Myocardial infarction or significant change in anginal pattern within one year prior to study entry or current congestive heart failure (New York Heart Association Class 2 or higher)
4. Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
5. History of invasive malignancy within the last five years prior to study entry except for carcinoma in situ or nonmelanoma skin cancer.
6. Psychiatric conditions which would prevent compliance with treatment or adequate informed consent.
7. Patients receiving another investigational agent during chemo- and radiotherapy
8. Uncontrolled intercurrent illness or other conditions that limit compliance with protocol treatment

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-08; Primary Completion 2010-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young Whang, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00225420?term=LCCC0420&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with high-risk or locally advanced prostate cancer were recruited from 2 institutions between December 2005 and January 2010.
Pre-assignment Details: Two patients were taken off the study due illness, two were removed because they were too large for the equipment, and one was removed due to CT screen failure.18 men with high-risk or locally advanced prostate cancer were enrolled. All 18 patients completed their radiation therapy and 16 completed all planned chemotherapy doses.
Groups:
- Docetaxel 10 mg/m2: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 10 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg intramuscular (IM) and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 centigray (cGy) in 200 cGy per fraction for a total of 39 treatments.
- Docetaxel 15 mg/m2: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 15 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg intramuscular (IM) and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments
- Docetaxel 20 mg/m2: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 20 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg intramuscular (IM) and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments
Period: Overall Study
Arm/Group | Docetaxel 10 mg/m2 | Docetaxel 15 mg/m2 | Docetaxel 20 mg/m2
Started | 9 | 6 | 3
Completed | 9 | 6 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included in this trial were high-risk localized (Gleason 8-10 or PSA level >= 20 ng/mL) prostate cancer, or T3 disease.
Groups:
- Overall Study: Single Arm Docetaxel: Docetaxel will be administered per the designated cohort starting at 10, 15 or 20 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg IM and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments.
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 62 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Clinical Stage [Count of Participants; unit: Participants] — The Classification of Malignant Tumours (TNM) system is a widely used cancer staging system. The T refers to the size and extent of the main tumor. The main tumor is usually called the primary tumor. T0 means the main tumor cannot be found. The higher the number following T, the larger the tumor or the more it has grown.
  Participants
    T1c-T2a | 9
    T2b-T2c | 5
    T3 | 4
Gleason Score [Count of Participants; unit: Participants] — A Gleason score is given based on how the prostate cancer tissue looks under the microscope. Gleason scores range from 2 to 10 and indicates how likely the tumor will spread. The higher the Gleason score the more likely the cancer tissue will spread.
  Participants
    Grade 7 | 3
    Grade 8-10 | 15
PSA level, ng/mL [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein produced by cells of the prostate gland. The PSA test measures the level of PSA in the blood. PSA levels are often elevated in men with prostate cancer.
  Participants
    <10 ng/mL | 6
    10-19 ng/mL | 4
    20-100 ng/mL | 5
    >100 ng/mL | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Dose-Limiting Toxicities
Description: Determine the number of patients experiencing dose-limiting toxicities (DLT) at each dose level. DLT was defined as grade 3-4 non-haematological or grade 4 haematological toxicity, using the Common Terminology Criteria for Adverse Events, version 3.0.
Time Frame: Average follow up of 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Docetaxel at 10 mg/m2: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 10 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg IM and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments.
- Docetaxel 15 mg/m2: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 15 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg IM and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments
- Docetaxel 20 mg/m2: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 20 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg IM and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments
Arm/Group | Docetaxel at 10 mg/m2 | Docetaxel 15 mg/m2 | Docetaxel 20 mg/m2
Number analyzed (Participants) | 9 | 6 | 3
Participants | 1 | 1 | 0

2. Secondary Outcome: Biochemical Progression-free Survival (PFS)
Description: Measure of the activity of a treatment on a disease. In this study it is measured from the date of enrollment to the date on which the prostate cancer progresses or the date the patient dies. Survival curves were estimated using the Kaplan-Meier technique. Biochemical (PSA) failure is defined, in accordance to the American Society for Therapeutic Radiology and Oncology consensus definition, as three consecutive rise in PSA. The date of biochemical failure is considered to be the midpoint between the last non-rising PSA and the first rising PSA.
Time Frame: Average follow up of 2 years
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Groups:
- Single Arm: Single Arm
  docetaxel: Docetaxel will be administered per the designated cohort starting at 10 mg/m2 intravenously over 1 hour weekly for eight weeks, for a total of eight treatments.
  leuprolide acetate: Leuprolide acetate will be administered at 22.5 mg IM and will be initiated 2 to 3 months prior to radiotherapy and chemotherapy with docetaxel.
  radiation therapy: The total dose will be 7800 cGy in 200 cGy per fraction for a total of 39 treatments.
Arm/Group | Single Arm
Number analyzed (Participants) | 18
percentage of patients | 94 [65 to 99]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=18)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4
Alkaline phosphatase (Investigations) | 4
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1
Bladder spasms (Renal and urinary disorders) | 1
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1 — decreased red blood cells
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Constitutional Symptoms (Other, specify) (General disorders) | 1 — Cold sensitivity
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 1
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3 — Fungal infection
Diarrhea (Gastrointestinal disorders) | 8
Distension/bloating, abdominal (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 4
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Edema: head and neck (General disorders) | 1
Edema: limb (General disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 11
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flu-like syndrome (General disorders) | 1
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 1 — Gastroesophageal reflux disease (GERD).
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 12
Hemorrhage, GI - Abdomen NOS (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 3
Hot flashes/flushes (Endocrine disorders) | 10
Hypertension (Cardiac disorders) | 5
Incontinence, anal (Gastrointestinal disorders) | 1
Infection - Other (Specify, __) (Infections and infestations) | 1 — Cold Symptoms
Insomnia (Psychiatric disorders) | 7
Leukocytes (total WBC) (Investigations) | 4
Libido (Reproductive system and breast disorders) | 1
Lymphopenia (Investigations) | 12
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 5
Mood alteration - Anxiety (Psychiatric disorders) | 2
Mood alteration - Depression (Psychiatric disorders) | 1
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 2 — leg cramps
Nausea (Gastrointestinal disorders) | 6
Neuropathy: sensory (Nervous system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Bladder (Renal and urinary disorders) | 1
Pain - Chest/thorax NOS (Cardiac disorders) | 1
Pain - Head/headache (Nervous system disorders) | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Pain - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 — Left shoulder
Pain - Penis (Reproductive system and breast disorders) | 1
Pain - Rectum (Gastrointestinal disorders) | 1
Pain - Stomach (Gastrointestinal disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Platelets (Investigations) | 6
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2 — Cold/upper respiratory infection
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 6 — Dysuria; painful urination; intermittent bladder spasms
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 2
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1
Ulcer, GI - Anus (Gastrointestinal disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 14
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2
Vasovagal episode (Nervous system disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight gain (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days